CLINICAL TRIAL: NCT04319055
Title: Artificial Intelligence-Assisted Facial, Periocular, and Orbital Analysis and Surgical Planning
Brief Title: AI-Assisted Facial Surgical Planning
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: 201908066RIND
Record Dates: First submitted 2020-03-03; First posted 2020-03-24 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Facial Plastic and Reconstructive Surgery; Periocular Diseases; Orbital Diseases; Artificial Intelligence
Keywords: Facial Plastic and Reconstructive Surgery; Periocular Diseases; Orbital Diseases; Artificial Intelligence
MeSH Terms: conditions — Orbital Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Computer vision using deep learning architecture is broadly used in auto-recognition. In the research, the deep learning model which is trained by categorized single-eye images is applied to achieve the good performance of the model in blepharoptosis auto-diagnosis.

DETAILED DESCRIPTION:
This auto-diagnosis system of blepharoptosis using machine learning architecture will assist in telemedicine, such as early screening of childhood ptosis for prompt referral and treatment. People could use this software via mobile devices to get a primitive diagnosis before they reach the physicians. Furthermore, in primary health care, where there is no oculoplastic surgeon, the software could assist primary care physicians or general ophthalmologists, in identifying the need for a referral.

ELIGIBILITY:
[Inclusion Criteria]

1. The participants who were 20-year-old or above,
2. Surgical informed consent was endorsed by the participants themselves,
3. Participants who have surgical indications of the oculofacial surgeries, and
4. The participants who agreed on photograph taking after explanation by the surgeon at outpatient clinics.

[Exclusion Criteria]

1. The participants who were 19-year-old or under,
2. The participants who don't have surgical indications of the oculofacial surgeries,
3. The participants who were designed for minimal invasive treatments, such as Botox or any kind of fillers injection,
4. The participants who refused photograph taking for any reason, and
5. The participants who are not available for standard quality of photograph taking, such as bedridden patients.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All data was collected at ophthalmic outpatient clinics of National Taiwan University Hospital.
Sampling Method: Probability Sample
Enrollment: 17932 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
The model performance is evaluated by accuracy | Through study completion, an average of 1 year
  An Artificial Intelligence Approach
AUC (Area Under the Curve) | Through study completion, an average of 1 year
  An Artificial Intelligence Approach
ROC (Receiver Operating Characteristics) curve. | Through study completion, an average of 1 year
  An Artificial Intelligence Approach
An Artificial Intelligence Approach to Identifying Facial, Periocular, and Orbital Diseases | Through study completion, an average of 1 year
  The model interpretability is accessed by Grad-CAM (Class Activation Maps).

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Lang Liao, MD,MPH, EMBA, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No